CLINICAL TRIAL: NCT04782245
Title: Acute Reno-Cardiac Action of Dapagliflozin In Advanced Heart Failure Patients on Heart Transplant Waiting List: a Multicenter, Double-blind, Randomized Clinical Trial.
Brief Title: Acute Reno-Cardiac Action of Dapagliflozin In Advanced Heart Failure Patients on Heart Transplant Waiting List
Acronym: ARCADIA-HF
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: New recommandations
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69HCL20_1135; 2020-005713-40 (EudraCT Number)
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: End-stage Heart Failure
Keywords: End-stage heart failure,; Cardio-renal syndrome; Dapagliflozin
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group Daplagliflozin (Experimental)
  Interventions: Drug: Dapagliflozin 10mg
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg — The intervention group will receive, during 6 months, dapagliflozin per oral route at a dose of 10 mg once daily in addition to the optimal medical management based on current heart failure practice guidelines.
  Arms: Treatment group Daplagliflozin
Drug: Placebo — Patients randomized in the control group will receive during 6 months, placebo once daily per oral route, in addition to the optimal medical management based on current heart failure practice guidelines.
  Arms: Control group

SUMMARY:
In the DAPA-HF trial, the use of dapagliflozin, an inhibitor of sodium-glucose cotransporter 2 (SGLT2), reduced significantly the risk of worsening heart failure or death from cardiovascular causes compared to placebo among patients with heart failure (HF) and a reduced ejection fraction. This new drug offers a very potent and interesting therapeutic pathway since it reduces clinical congestion, it preserves glomerular renal function, does not appear to cause symptomatic clinical hypotension and improves symptoms and quality of life compared to placebo.

Advanced heart failure patients with reduced ejection fraction represent a small and severe subgroup of heart failure of patients with frequent worsening heart failure events and high rates of death. The effect of dapagliflozin in this subgroup of patients was not assessed in the DAPA-HF study. The therapeutic profile of SGLT2 inhibitors appears to be of high interest, since this group of patients has a poor tolerance to usual heart failure drugs, frequent worsening renal function and congestive symptoms persistence with poor quality of life scores.

Soluble urokinase-type plasminogen activator receptor (suPAR) is a signaling glycoprotein considered to be involved in the pathogenesis of kidney disease. It is associated with the risk of acute kidney injury in different clinical and experimental situation. It is also a new validated biomarker predictive of adverse clinical outcome in heart failure patients. This biomarker allows a better risk stratification in heart failure patients after adjustment for Nt-proBNP.

As a useful biomarker implicated in both heart failure and acute kidney injury, suPAR seems to be an interesting biomarker to assess cardio-renal benefits of dapagliflozin.

The aim of this study is to investigate if a treatment by dapagliflozin reduces significantly suPAR compared to placebo in a population of advanced heart failure patients, candidates to heart transplantation. The effect of dapagliflozin compared to placebo will also be assessed on other secondary heart failure outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed informed consent form
2. Age ≥ 18 years
3. NYHA class ≥3
4. LVEF ≤ 35%
5. On optimal medical management (OMM) based on current heart failure practice guidelines at maximal tolerated dose for at least 30 days
6. On waiting list for heart transplantation after multidisciplinary Heart Team decision, with anticipated access to heart transplant ≥ 6 months

Exclusion Criteria:

1. Priority patient on waiting list for heart transplantation
2. Etiology of heart failure due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis or restrictive cardiomyopathy
3. Inotrope dependent, existence of ongoing mechanical circulatory support
4. Current acute decompensated HF or hospitalization due to decompensated HF <30 days prior to the enrolment
5. History of any organ transplant or prior implantation of a ventricular assistance device (VAD) or similar device, or implantation expected after randomization
6. Presence of an active, uncontrolled infection
7. Any recent interventional procedure likely to improve symptoms and heart failure status (coronary revascularization, percutaneous mitral valve intervention, cardiac resynchronization therapy) < 60 days
8. Glomerular filtration rate < 30 ml/min/1.73 m2, according to CKD-EPI formula
9. Unstable or rapidly progressing renal disease
10. Patients with severe hepatic impairment (Child-Pugh class C)
11. Chronic treatment with dapagliflozin or other SGLT2 inhibitors
12. Patient with known history of severe drug intolerance to dapagliflozin or any excipients of the dapagliflozin (galactose, lactase)
13. Type 1 diabetes mellitus
14. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or extraction of study drug at investigators' discretion
15. Participation in another clinical interventional trial
16. Any condition other than heart failure that could limit survival to less than 24 months
17. Positive pregnancy test if of childbearing potential or refusal to use adequate contraception or women breast-feeding
18. Patients with any legal protection measure
19. Patients without any health coverage
20. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychological issues that are likely to impair compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Levels of suPAR (ng/ml) | 6 months

SECONDARY OUTCOMES:
VO2 max assessment | 6 months
  VO2 max assessment to evaluate the functional status
cardiac output assessed by right heart catheterization | 6 months
  The impact of dapagliflozin on hemodynamic parameters between baseline and 6 months assessed by right heart catheterization hemodynamic parameters
pulmonary capillary wedge pressure assessed by right heart catheterization | 6 months
  The impact of dapagliflozin on hemodynamic parameters between baseline and 6 months assessed by right heart catheterization hemodynamic parameters
pulmonary artery systolic and mean pressure assessed by right heart catheterization | 6 months
  The impact of dapagliflozin on hemodynamic parameters between baseline and 6 months assessed by right heart catheterization hemodynamic parameters
mean pressure assessed by right heart catheterization | 6 months
  The impact of dapagliflozin on hemodynamic parameters between baseline and 6 months assessed by right heart catheterization hemodynamic parameters
right atrial pressure assessed by right heart catheterization | 6 months
  The impact of dapagliflozin on hemodynamic parameters between baseline and 6 months assessed by right heart catheterization hemodynamic parameters
Left Ventricular Ejection Function assessed by echocardiography | 6 months
  The impact of dapagliflozin on echocardiographic parameters between baseline and 6 months
Left ventricular end-diastolic diameter assessed by echocardiography | 6 months
  The impact of dapagliflozin on echocardiographic parameters between baseline and 6 months
Left ventricular end systolic volume assessed by echocardiography | 6 months
  The impact of dapagliflozin on echocardiographic parameters between baseline and 6 months
mitral regurgitation grade assessed by echocardiography | 6 months
  The impact of dapagliflozin on echocardiographic parameters between baseline and 6 months
left atrial volume assessed by echocardiography | 6 months
  The impact of dapagliflozin on echocardiographic parameters between baseline and 6 months
Nt-proBNP level | 6 months
Creatinine level | 6 months
Quality of life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BAUDRY, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Pneumologique et Cardiovasculaire Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided